CLINICAL TRIAL: NCT02262858
Title: Bioequivalence of 80 mg Telmisartan/12.5 mg HCTZ Fixed Dose Combination Compared With Its Monocomponents in Healthy Male Volunteers II (an Open-label, Randomised, Single-dose, Two-sequence, Four-period Replicated Crossover Study)
Brief Title: Bioequivalence of Telmisartan/ HCTZ Fixed Dose Combination Compared With Its Monocomponents in Healthy Male Volunteers II
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 502.495
Record Dates: First submitted 2014-10-10; First posted 2014-10-13 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Telmisartan; Hydrochlorothiazide

ARMS (2):
- Telmisartan and HCTZ (fix dose combination) (Experimental)
  Interventions: Drug: Telmisartan and HCTZ
- Telmisartan and HCTZ (monocomponent) (Active Comparator)
  Interventions: Drug: Telmisartan; Drug: HCTZ

INTERVENTIONS:
Drug: Telmisartan and HCTZ
  Arms: Telmisartan and HCTZ (fix dose combination)
Drug: Telmisartan
  Arms: Telmisartan and HCTZ (monocomponent)
Drug: HCTZ
  Arms: Telmisartan and HCTZ (monocomponent)

SUMMARY:
Study to investigate the bioequivalence of 80 mg telmisartan/12.5 mg hydrochlorothiazide (HCTZ) fixed dose combination compared with its monocomponents

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males according to the following criteria:

   Based upon a complete medical history, physical finding, physical examination (measurements of height and body weight), vital signs (blood pressure, pulse rate), 12- lead ECG, clinical laboratory tests (including gastric acid (GA) test)
   * No finding of clinical relevance
   * No evidence of a clinically relevant concomitant disease
2. Age ≥ 20 years and Age ≤ 35 years
3. Body weight ≥ 50 kg
4. Body mass index (BMI) ≥ 17.6 kg/m2 and BMI ≤ 25.0 kg/m2
5. Signed and dated written informed consent prior to admission to the study

Exclusion Criteria:

1. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Surgery of gastrointestinal tract (except appendectomy)
3. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
4. History of relevant orthostatic hypotension, fainting spells or blackouts
5. Chronic or relevant acute infections
6. History of allergy/hypersensitivity (including drug allergy) which was deemed relevant to the trial as judged by the investigator
7. Positive result for hepatitis B surface antigen (HBsAg), anti hepatitis C virus (HCV), syphilitic test or human immunodeficiency virus (HIV) antigen-antibody test
8. Intake of drugs with a long half-life (≥ 24 hours) within at least 1 month prior to administration or within a period of 10 or less half-lives of the respective drugs during the trial
9. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
10. Participation in another trial with an investigational drug within 4 months prior to administration or during the trial
11. Smoker (20 or more cigarettes/day)
12. Inability to refrain from smoking during hospitalization
13. Alcohol abuse (60 g or more ethanol/day: ex. 3 middle-sized bottles of beer, 3 gous (equivalent to 540 mL) of sake)
14. Drug abuse
15. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
16. Excessive physical activities (within one week prior to administration or during the trial)
17. Any laboratory value outside the reference range that was of clinical relevance
18. Inability to comply with dietary regimen of study centre
19. Any other volunteers whom the investigator or sub investigator did not allow to participate in this study

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2005-08; Primary Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) | up to 72 hours after drug administration
Cmax (maximum measured concentration of the analyte in plasma) | up to 72 hours after drug administration

SECONDARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 72 hours after drug administration
tmax (time from dosing to the maximum concentration of the analyte in plasma) | up to 72 hours after drug administration
λz (terminal rate constant of the analyte in plasma) | up to 72 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 72 hours after drug administration
MRTpo (mean residence time of the analyte in the body after po administration) | up to 72 hours after drug administration
Number of subjects with adverse events | up to 7 days after last drug administration
Number of subjects with clinically significant changes in vital signs | up to 7 days after last drug administration
  blood pressure, pulse rate
Number of subjects with clinically significant changes in 12 lead ECG | up to 7 days after last drug administration
Number of subjects with clinically significant changes in laboratory tests | up to 7 days after last drug administration